CLINICAL TRIAL: NCT05556109
Title: Possible Role of Inflammatory Serum Biomarkers in Differentiation Between Epileptic Seizure and Psychogenic Non-epileptic Seizure
Brief Title: Inflammatory Biomarkers in Seizure
Acronym: seizure
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Mostafa Ahmed Abdel Aal, Doctor, Assiut University
Other Study IDs: Biomarkers in seiz
Record Dates: First submitted 2022-09-23; First posted 2022-09-27 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Biomarkers in Seizures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Epileptic seizure: patients diagnosed as epileptic seizure are aged >12 years
  Interventions: Diagnostic Test: Inflammatory serum biomarkers
- Psychogenic non-epileptic seizure: patients diagnosed as psychogenic non-epileptic seizure are aged >12 years
  Interventions: Diagnostic Test: Inflammatory serum biomarkers
- Normal healthy control: Heathy control are aged >12 years with no history of lifetime seizures or suspected seizures or febrile seizure and no treatment with an antiepileptic drug (AED) prior to blood draw
  Interventions: Diagnostic Test: Inflammatory serum biomarkers

INTERVENTIONS:
Diagnostic Test: Inflammatory serum biomarkers — Measuring inflammatory serum biomarkers by ELISA

SUMMARY:
1. Evaluation of the role of TRAIL and MCP-2 in differentiation between epileptic seizure and psychogenic non-epileptic seizure.
2. Possible role to predict the prognosis of patients with epileptic seizure

DETAILED DESCRIPTION:
Epilepsy is one of the most prevalent neurological disorders characterized by frequent somatic and psychiatric co-morbidities(1). Accurate diagnosis of epilepsy is challenging because clinicians rarely observe the actual clinical seizure outside of the hospital. Furthermore, psychogenic nonepileptic seizures (PNES) can mimic epileptic seizures (ES), leading to erroneous diagnosis and inappropriate treatments. A critical gap in the diagnostic assessment of seizures is a blood test that can distinguish ES from PNES (2). Both diagnoses were confirmed by the gold standard diagnostic method video/electroencephalogram (EEG) monitoring (3). Taking all in to account, the notion that neuro-inflammation is the key pathology behind focal epileptic seizure initiation and maintenance and the dynamic and adaptative process of neuro -inflammation is associated with blood-brain-barrier disruption and glial activation is no longer a surprise (4).

Tumor necrosis factor related apoptosis inducing ligand (TRAIL) regulates immune responses via apoptosis, with lower levels associated with severe infection, including sepsis (5). Monocyte chemoattractant protein-2 (MCP-2) has been well recognized to participate in immune regulation via binding to chemokine receptors and activation chemotaxis in lymphocytes T, natural killer (NK) cells, and monocytes therefore contributing to the pathogenesis of monocyte-dependent tissue injury (6). Hence, MCP-2 overexpression could result in an increased immune response. Further, since increased levels of MCP-2 have been observed in patients with Alzheimer's disease, this may further support the existence of the biodirections relationship between neurodegeneration and seizures/epilepsy (7).

ELIGIBILITY:
Inclusion Criteria:

patients diagnosed as epileptic seizure are aged >12 years patients diagnosed as psychogenic non-epileptic seizure are aged >12 years Normal healthy control for comparison. Heathy control are aged >12 years with no history of lifetime seizures or suspected seizures or febrile seizure and no treatment with an antiepileptic drug (AED) prior to blood draw

Exclusion Criteria:

* Neurological criteria: Other CNS disorders including Parkinson's disease, amyotrophic lateral sclerosis ,cerebrovascular stroke, Psychiatric disorders {major depression disorder , generalized anxiety, mania and other psychiatric diseases).

Others: Tumors and cardiovascular

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients diagnosed as epileptic seizure are aged >12 years patients diagnosed as psychogenic non-epileptic seizure are aged >12 years Normal healthy control for comparison. Heathy control are aged >12 years with no history of lifetime seizures or suspected seizures or febrile seizure and no treatment with an antiepileptic drug (AED) prior to blood draw
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Detection of the level of inflammatory biomarkers in epileptic seizure and psychogenic non-epileptic seizure | 2 years
  Evaluation of the role of TRAIL and MCP-2 in differentiation between epileptic seizure and psychogenic non-epileptic seizure